CLINICAL TRIAL: NCT02254785
Title: A Phase II, Randomized, Multi-center Study of Cabazitaxel Versus Abiraterone or Enzalutamide in Poor Prognosis-metastatic Castration-resistant Prostate Cancer
Brief Title: Cabazitaxel vs Abiraterone or Enzalutamide in Patients With Poor Prognosis Metastatic Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Sanofi (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZM-054
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Castration-Resistant Prostatic Cancer
Keywords: poor prognosis; castrate-resistant prostate cancer; cabazitaxel; abiraterone; enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — cabazitaxel; abiraterone; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabazitaxel (Experimental)
  Interventions: Drug: cabazitaxel
- Abiraterone or enzalutamide (Active Comparator)
  Interventions: Drug: Abiraterone; Drug: Enzalutamide 160mg daily (oral)

INTERVENTIONS:
Drug: cabazitaxel — Cabazitaxel 25mg/m2 intravenous every 3 weeks until disease progression
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: Abiraterone — Abiraterone 1000mg daily (oral) until disease progression
  Other Names: Zytiga
  Arms: Abiraterone or enzalutamide
Drug: Enzalutamide 160mg daily (oral) — Enzalutamide 160mg daily (oral) until disease progression
  Other Names: Xtandi
  Arms: Abiraterone or enzalutamide

SUMMARY:
The purpose of this study is to assess and compare the clinical benefit rate in patients with metastatic castrate-resistant prostate cancer and poor prognostic factors treated with cabazitaxel or novel hormonal agents (abiraterone or enzalutamide) as initial therapy, to determine which treatment is most active in this population. Clinical benefit rate is defined as PSA or measurable radiological response of any duration or stable disease for > or equal to 12 weeks, in the absence of other indicators of progression.

There is option to cross-over onto the other arm if the patient progresses.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate adenocarcinoma.
* Able and willing to provide informed consent and to comply with the study procedures
* Age ≥18
* Evidence of metastatic disease on a chest, abdominal, or pelvic CT scan and/or bone scan within 6 weeks of registration
* Castration resistant disease defined as evidence of radiological and/or PSA progression despite castrate levels of testosterone (serum testosterone < 50 ng/dL (1.7 nmol/L)). For PSA progression, there must be at least 2 sequential rises at a minimum of 1-week intervals. The first PSA value must be ≥ 2. (Prostate Cancer Working Group 2 (PCWG2) criteria)
* Poor prognosis disease as defined by any of the following:

the presence of liver metastases OR development of castration-resistance within 12 months of orchiectomy or commencement of LHRH antagonist/agonist for metastatic disease OR the presence of 4 or more of the following factors:

* LDH > ULN
* ECOG Performance status (PS) 2
* visceral metastatic disease
* serum albumin less than or equal to 4 g/dL
* ALP > ULN
* or < 36 months from commencement of initial androgen deprivation therapy to study enrollment
* ECOG PS 0-2.
* Adequate end-organ function within 14 days of registration:

Haemoglobin ≥ 90 g/L Neutrophils ≥ 1.5 x 109 /L Platelets ≥ 100 x 109/L AST < 1.5 x ULN ALT < 1.5 x ULN Bilirubin ≤ 1.0 x ULN (exceptions for Gilbert's syndrome) Creatinine ≤ 1.5 x ULN

* At least 21 days have passed since completing radiotherapy (exception for radiotherapy: at least 7 days since completing a single fraction of ≤ 800 cGy to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit) at the time of randomization.
* At least 21 days have passed since receiving any investigational agent at the time of registration.
* At least 21 days have passed since major surgery.
* Neuropathy ≤ grade 1 at the time of registration.
* Has recovered from all therapy-related toxicity to ≤ grade 2 (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy) at the time of registration.
* Eligible for abiraterone acetate and/or enzalutamide as per standard of care practices.

Exclusion Criteria:

* Histologic evidence of small cell/neuroendocrine prostate cancer.
* Other chemotherapy regimen beyond one prior course of docetaxel.
* Previously received treatment with cabazitaxel.
* Received any prior next-generation anti-androgen (e.g. enzalutamide, ARN-509) or CYP 17 inhibitors (e.g. abiraterone, TAK-700).
* Other condition, illness, psychiatric condition, or laboratory abnormality that may increase the risk associated with administration of cabazitaxel, abiraterone or enzalutamide, study participation, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate | 12 weeks or more
  To assess and compare the clinical benefit rate in patients with mCRPC and poor prognostic factors treated with cabazitaxel or novel hormonal agents (abiraterone or enzalutamide) as initial therapy, to determine which treatment is most active in this population. Clinical benefit rate is defined as PSA or measurable radiological response of any duration or stable disease for greater than or equal to 12 weeks, in the absence of other indicators of progression.

SECONDARY OUTCOMES:
Duration of treatment time to progression | 12 weeks until disease progression
  To measure the treatment time before any type of progression (symptomatic, PSA, or radiological) between Arm A and Arm B
Progression Free Survival | 12 weeks until disease progression
  To measure the progression-free survival of metastatic castration-resistant prostate cancer patients following treatment with cabazitaxel or abiraterone/enzalutamide as initial therapy.
Overall Survival | 12 weeks until 2 years after last study visit
  To measure the overall survival of metastatic castration-resistant prostate cancer patients following treatment with cabazitaxel or abiraterone/enzalutamide as initial therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Principal Investigator — British Columbia Cancer Agency
Locations (15):
- Australia (3):
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health-Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (12):
  - Tom Baker Cancer Cantre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA- Vancouver Center, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Durham Regional Cancer Centre (Lakeridge Health), Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Annala M, Fu S, Bacon JVW, Sipola J, Iqbal N, Ferrario C, Ong M, Wadhwa D, Hotte SJ, Lo G, Tran B, Wood LA, Gingerich JR, North SA, Pezaro CJ, Ruether JD, Sridhar SS, Kallio HML, Khalaf DJ, Wong A, Beja K, Schonlau E, Taavitsainen S, Nykter M, Vandekerkhove G, Azad AA, Wyatt AW, Chi KN. Cabazitaxel versus abiraterone or enzalutamide in poor prognosis metastatic castration-resistant prostate cancer: a multicentre, randomised, open-label, phase II trial. Ann Oncol. 2021 Jul;32(7):896-905. doi: 10.1016/j.annonc.2021.03.205. Epub 2021 Apr 6. PMID 33836265